CLINICAL TRIAL: NCT04995107
Title: Effectiveness of Electro-Press Needle for Menopause-associated Hot Flashes: Protocol of a Randomized Controlled Trial
Brief Title: Effectiveness of Electro-Press Needle for Menopause-associated Hot Flashes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yu Shudan, principal investigator,resident doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-047-KY-01
Record Dates: First submitted 2021-08-01; First posted 2021-08-06 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Hot Flashes; Acupuncture Therapy; Perimenopausal Disorder; Postmenopausal Symptoms
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statisticians and outcome assessors will be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-Press Needle group (Experimental): Body acupoints of Yintang (GV29), Dazhui (GV14), Guanyuan (CV4), bilateral Zigong (EX-CA1), and bilateral Sanyinjiao (SP6) and auricular acupoints of Heart (CO15), Chuiqian (LO4) and Shenmen (TF4) will be selected for treatment. Auricular acupoints on right and left ear will be stimulated alternatively, one side on each time.The treatment will last 40mins for each session, 3 sessions a week (ideally every other day) for a succession of 6 weeks.
  Interventions: Device: Electro Press needle
- Waiting-list group (No Intervention): Participants in the waiting-list group will receive no intervention for 6 weeks and be followed up till weeks 30.

INTERVENTIONS:
Device: Electro Press needle — Body acupoints will be stimulated by the press needles 0.25mm in diameter and 2mm in length and ear acupoints will be stimulated by the press needles 0.25mm in diameter and 0.9mm in length (all from ZhenXing Brand, Hangzhou Yuanli Medical Appliance Factory, China). After sterilization of the local skin, the needle will be pressed to the acupoints and the tape will be sticked to the skin. Then, the electric device (φ44×15.8mm Type ZXHPAMDZB-02C) together with the electrode patch will be sticked to the surface of skin (on top of the sticky tapes of the press needle) in the area of CV4 and bilateral EX-CA1, and bilateral SP6 respectively. The electric device will be switch to the mode of "dense intermittent wave", and the current intensity will be increased gradually till the muscles around jumps slightly.All the needles on the body acupoints will be removed after each session, while those on the auricular acupoints can be kept for as long as 6 hours (removed before going to bed).
  Other Names: EPN
  Arms: Electro-Press Needle group

SUMMARY:
The investigators plan to conduct the randomized controlled trial to evaluate the effectiveness of electro-press needle (EPN), a novel acupuncture needle combining shallow and gentle insertion with transdermal electrical stimulation, on menopause-associated hot flash in comparison with waiting-list group among women during menopausal transition and postmenopausal periods.

DETAILED DESCRIPTION:
As the most common type of menopause-associated symptoms, hot flashes affect up to 85% of women aging between 40 and 65 years . In China, women suffer from hot flushes as long as 4 to 5 years on average, some of whom may bear the symptoms for 12 years.Hormone replacement therapy (HRT) is generally recommended to relieve menopause-associated hot flashes.However, long-term usage of HRT may increase the incidence of endometrial, breast and ovarian cancer, thrombosis and strokes.Results of previous studies indicated that acupuncture might help to relieve the symptoms.There is insufficient evidence supporting its effectiveness for relieving the hot flash symptom.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 40-60 years old;
2. Scoring 14 points or more in at least one day during the one-week baseline assessment, or having an average of ≥ 7 moderate or severe heating per 24 hours recorded in HF Dairy ;
3. Fulfilling either condition mentioned below:

   1. The last menstrual period was more than 12 months ago (including 12 months);
   2. In the late menopausal transition, and has amenorrhea for more than 60 days;
   3. FSH≥25IU, and has vasomotor symptoms of HF, sweating, insomnia, migraine, or restlessness, etc.
4. Volunteer to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Usage of HRT via transdermal administration in the previous one month, or via oral or intrauterine administration in the previous two months; usage of phytoestrogens therapy, transvaginal estrogen administration, or estrogen or progesterone injections in the previous three months;
2. Bilateral salpingo-oophorectomy;
3. Amenorrhea secondary to premature ovarian failure, ovarian cyst or tumor, thyroid disease, hyperprolactinemia, or Cushing's syndrome, etc.;
4. Accepted acupuncture or drugs to treat the symptoms of HF within the previous 3 months;
5. Received radiotherapy or chemotherapy before;
6. Coagulation dysfunction, or taking warfarin, heparin and other anticoagulant drugs at present;
7. Suffering from skin diseases, such as eczema, psoriasis, etc.;
8. Severe hepatic and renal insufficiency;
9. Uncontrolled hypertension, diabetes or thyroid disease;
10. Diabetic neuropathy and mental illness (including depression);
11. Being pregnant, breastfeeding or planning to be pregnant during the trial;
12. Regular usage of sedatives or anti-anxiety drugs;
13. Smoking for more than 5 years (at least twenty cigarettes a day on average) , or with the problem of alcohol abuse;
14. Installation of pacemakers;
15. Poor compliance.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 122 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with a reduction of 50% or more on the mean 24-hour HF score from baseline | week 6
  The mean 24-hour HF score = (1 × number of mild HF + 2 × number of moderate HF + 3 × number of severe HF + 4 × number of very severe HF)/Number of days reported.

SECONDARY OUTCOMES:
The proportion of participants with a reduction of 50% or more on the mean 24-hour HF score from baseline | week 3,18,30
  The mean 24-hour HF score = (1 × number of mild HF + 2 × number of moderate HF + 3 × number of severe HF + 4 × number of very severe HF)/Number of days reported.
The proportion of participants with a reduction of 50% or more in the mean 24-hour HF frequency from baseline | week 3,6,18,30
  The mean 24-hour HF frequency = total number of HF reported/Number of days reported.
The proportion of patients with at least a 50% reduction in the mean 24-hour HF severity from baseline | week 3,6,18,30
  The mean 24-hour HF severity = (1 × number of mild HF + 2 × number of moderate HF + 3 × number of severe HF + 4 × number of very severe HF)/ Number of HF reported.
The changes in the mean 24-h HF score from baseline | week 3,6,18,30
  The mean 24-hour HF score = (1 × number of mild HF + 2 × number of moderate HF + 3 × number of severe HF + 4 × number of very severe HF)/Number of days reported.
The change of Menopause rating scale (MRS) score from baseline | week6, 18 and 30
  MRS is a common menopause specific subscale, including 11 items from psychological, somatic to urogenital, with 5 as minimal clinically important differences(MCID).
TThe change of Menopause-Specific Quality of Life Questionnaire (MENQOL) score from baseline | week 6, 18 and 30
  MENQOL consists of 29 items assessing four domains: VMS, physical symptoms, psychological symptoms, and urogenital/sexual symptoms,with 4 as minimal clinically important differences(MCID).
The proportion of participants reporting "significantly reduced" or "moderately reduced" based on Global Response Assessment (GRA) | week 3 ,6, 18 and 30
  The response of participants to the treatments are divided into seven grades by GRA: significantly reduced, moderately reduced, slightly reduced, no change, slightly aggravated, moderately aggravated and significantly aggravated. The proportion of participants reporting "significantly reduced" or "moderately reduced" are recorded as the response rate of the overall efficacy.

OTHER OUTCOMES:
Participants'acceptability towards EPN | week 1 and 3,at the end of the first and ninth treatments
  Use the 3-point method to evaluate, unacceptable (0 points), acceptable (1 points), easy to accept (2 points), patients who cannot accept should be written the reason clearly.Only patients in electric press needle group will score.
Participants' belief that EPN might help | Baseline assessmentweek 0
  Participants in the EPN group will answer the following question before the first intervention: "Do you think acupuncture will be effective for treating the disease?"The participants can answer "Yes", "No", or "Unclear."
Participants' expectations of improvement to menopausal associated hot flashes | Baseline assessment week 0
  Participants in the EPN group will answer the following question before the first intervention: "Do you think acupuncture will be effective for improving menopausal associated HF?" The participants can answer "Yes", "No", or "Unclear."
Safety assessment | Through study completion
  Adverse events and severe adverse events will be recorded in case report form, whether related to interventions or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Acupuncture, Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the article after deidentification, excluding the private information of participants.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning immediately after publication and ending 6 months following article publication
Access Criteria: Proposals should be directed to miaomiao101@126.com. To gain access, data requestors wil need to sign a data access agreement.

REFERENCES:
- [Derived] Yu S, He X, Shi H, Chen Y, Liu Z. Effectiveness of electro-press needle for menopause-associated hot flashes: Protocol of a randomized controlled trial. Medicine (Baltimore). 2022 Feb 11;101(6):e28597. doi: 10.1097/MD.0000000000028597. PMID 35147087